CLINICAL TRIAL: NCT01951027
Title: A Dose-block Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Study to Investigate the Safety, Tolerability, and PK/PD of GX-G3 After Single SC Administration in Healthy Male Subjects
Brief Title: Phase I Study GX-G3 in Healthy Subjects
Acronym: GX-G3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: GX-G3_HV_1
Record Dates: First submitted 2013-09-17; First posted 2013-09-26 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics; Pharmacodynamics; DLT; Immunogenecity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): GX-G3 12.5 μg/kg or Placebo
  Interventions: Drug: GX-G3 12.5 μg/kg or Placebo
- Cohort 2 (Experimental): GX-G3 25 μg/kg or Placebo
  Interventions: Drug: GX-G3 25 μg/kg or Placebo
- Cohort 3 (Experimental): GX-G3 50 μg/kg or Placebo
  Interventions: Drug: GX-G3 50 μg/kg or Placebo
- Cohort 4 (Experimental): GX-G3 100 μg/kg or Placebo
  Interventions: Drug: GX-G3 100 μg/kg or Placebo

INTERVENTIONS:
Drug: GX-G3 12.5 μg/kg or Placebo — Single SC injection
  Other Names: GX-G3(G-CSF-hyFc)
  Arms: Cohort 1
Drug: GX-G3 25 μg/kg or Placebo — Single SC injection
  Other Names: GX-G3(G-CSF-hyFc)
  Arms: Cohort 2
Drug: GX-G3 50 μg/kg or Placebo — Single SC injection
  Other Names: GX-G3(G-CSF-hyFc)
  Arms: Cohort 3
Drug: GX-G3 100 μg/kg or Placebo — Single SC injection
  Other Names: GX-G3(G-CSF-hyFc)
  Arms: Cohort 4

SUMMARY:
pharmacokinetics/pharmacodynamics of GX-G3 after single subcutaneous administration in healthy male subjects.

DETAILED DESCRIPTION:
MTD will be determined by DLT occurrence and frequency, and severity and charactoristic of adverse event, vital sign, physical examination, ECG, Laboratory test, chest-X-ray will be examined for safety evaluation.

The second purpose is to evaluate pharmacokinetics and pharmacodynamics, and immunogenecity will be evaluated to investigate antibody production.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be entered in the study only if they meet all of the following criteria:

1. Are capable of understanding and complying with the requirements of the study and have voluntarily signed the informed consent form (ICF);
2. Healthy male volunteers aged 20-45 years;
3. Have a body weight of 60-90 kg (inclusive), have a body mass index (BMI) equal to or greater than 19 and less than 27 kg/m2;
4. Are eligible for the study based on screening data (Subjects may participate if Investigator considered eligible after looking at other screening data);

Exclusion Criteria:

Subjects presenting with any of the following will not be entered in to the study:

1. Have a history of or current evidence of disease;
2. Have percent of white blood cell (WBC) or neutrophil > UNL;
3. Have count of platelet < 100,000/mm3;
4. Have the longest length of spleen > 16 cm measured by abdomen ultrasonography ;
5. Have MSSBP ≥ 140 mmHg or ≤ 90 mmHg and/or MSDBP ≥ 95 mmHg or ≤ 50 mmHg; (BP must be measured after resting for at least 3 minutes)
6. Have clinically significant arrhythmia by EKG/ECG;
7. Are positive for HBV, HCV, HIV;
8. Have a history of allergy/hypersensitivity or ongoing allergy/hypersensitivity to any drug, as judged by the investigator;
9. Have had any blood donation/ blood loss greater than 400 ml within 8 weeks prior to dosing;
10. Have participated in another clinical trial with investigational drugs within 8 weeks of screening period;
11. Any other conditions that are considered inappropriate or unsafe for subjects by the Investigator;
12. Are considered ineligible by the investigator due to physical findings or laboratory values at the screening assessments;
13. Have a history of G-CSF treatment;

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
DLT incidence and frequency after GX-G3 single S.C. injection | 6 weeks
  [DLT criteria: CTCAE V4.03]
  1. Hematologic type: grade 3 Hematologic N.O.S, grade 3 or 4 Leukocytosis
  2. Non-Hematologic: grade 3 N.O.S
     * N.O.S: not otherwise specified
     * Leukocytosis: continued more than 5 days, grade 3(>100,000 cells/mm3), or grade 4(clinical manifestations of leucostasis; urgent intervention indicated)

SECONDARY OUTCOMES:
Adverse events incidence and frequency at each dose group after GX-G3 single injection | 6 weeks
Pharmacokinetics parameters after GX-G3 single injection | 3 weeks
  AUC/D, Cmax/D, AUC, AUClast, Cmax, tmax, half-life
Pharmacodynamics parameters after GX-G3 single injection | 3 weeks
  Emax, Emax, Tmax and AUEClast of absolute neutrophil count(ANC), WBC count and CD34+ cell count

CONTACTS AND LOCATIONS:
Overall Officials: Sang-In Yang, Ph.D, Study Director — Genexine, Inc, Clinical development Department; Jae Woo Kim, M.D., Principal Investigator — CHUNGNAM NATIONAL UNIVERSITY HOSPITAL Clinical Research Center
Locations (1):
- Chungnam National University Hospital, Jung-gu, Daejeon, South Korea